CLINICAL TRIAL: NCT01447095
Title: Effect of Prostacyclin Infusion on Cerebral Vessels, Cerebral Bloodflow and Cerebral Metabolism in Patients With Subarachnoid Haemorrhage
Brief Title: Effects of Prostacyclin Infusion on Cerebral Vessels and Metabolism in Patients With Subarachnoid Haemorrhage
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rune Rasmussen (Other)
Responsible Party: Sponsor-Investigator, Rune Rasmussen, MD, Sponsor-Investigator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2011-002798-50
Record Dates: First submitted 2011-10-02; First posted 2011-10-05 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Subarachnoid Hemorrhage
Keywords: Subarachnoid hemorrhage; vasospasm; prostacyclin
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Epoprostenol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low dose prostacyclin (Active Comparator)
  Interventions: Drug: Prostacyclin 1 ng/kg/min
- High dose prostacyclin (Active Comparator)
  Interventions: Drug: Prostacyclin 2 ng/kg/min
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prostacyclin 1 ng/kg/min — Continuous i.v. infusion of epoprostenol 1 ng/kg/min day 5-10 after SAH
  Other Names: Flolan
  Arms: Low dose prostacyclin
Drug: Prostacyclin 2 ng/kg/min — Continuous i.v. infusion of epoprostenol 2 ng/kg/min day 5-10 after SAH
  Other Names: Flolan
  Arms: High dose prostacyclin
Drug: Placebo — Continuous i.v. infusion with placebo day 5-10 after SAH
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether prostacyclin is effective in prevention of cerebral vasospasm in patients with subarachnoidal hemorrhage (SAH).

ELIGIBILITY:
Inclusion Criteria:

* SAH verified by CT
* Aneurysm identified and treated
* Fisher grade 3 + 4
* WFNS grade 1-4 (World Federation of Neurosurgical Societies )

Exclusion Criteria:

* Pregnancy/lactation
* Heard failure
* Kidney failure
* Liver failure
* Hemorrhagic diathesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Radiographic vasospasm measured by CT perfusion | Day 8 (+/- 1 day) after aneurysm treatment
  Changes in regional cerebral blood flow from baseline in the arterial territories of the anterior cerebral artery, medial cerebral artery and the posterior cerebral artery

SECONDARY OUTCOMES:
Cerebral metabolism measured by microdialysis | every 2. hour day 3-10 after aneurysm treatment
  Cerebral metabolism measured by microdialysis. Lactate, pyruvate, glucose, glutamate and glycerol are measured.
Glasgow outcome scale (GOS) at 3 months | 3 months efter SAH
  Glasgow outcome scale (GOS) at 3 months obtained by telephone interview.
Clinical vasospasm | day 5-10 after SAH
  Clinical vasospasm defined as delayed neurological deficits (DIND).
Brain tissue oxygen (PtiO2) | continuous measurement day 3-10 after SAH
  Brain tissue oxygen (PtiO2) measured by Licox catheter.
Mean arterial pressure (MAP) | Continuous day 1-10 after SAH
  Mean arterial pressure (MAP) measured by arterial catheter.
Radiographic vasospasm measured by CT angiography | Measured day 8 +/- 1 day
  Qualitative assessment (none, mild/moderate, severe) of vasospasm.
Level of brain damage biomarker | daily day 4-11 after SAH
  Serum levels of S100b in peripheral blood

OTHER OUTCOMES:
Neuropeptide Y | May 2014
  Neuropeptide Y will be measured in all patients Day 2-11. The concentration will be related to CBF, angiographic vasospasm and clinical outcome for all patients. The results will be reported in a separate puplication.

CONTACTS AND LOCATIONS:
Overall Officials: Rune Rasmussen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, dep. of neurosurgery, Copenhagen, Denmark

REFERENCES:
- [Derived] Rasmussen R, Wetterslev J, Stavngaard T, Juhler M, Skjoth-Rasmussen J, Grande PO, Olsen NV. Effects of prostacyclin on cerebral blood flow and vasospasm after subarachnoid hemorrhage: randomized, pilot trial. Stroke. 2015 Jan;46(1):37-41. doi: 10.1161/STROKEAHA.114.007470. Epub 2014 Nov 20. PMID 25414173
- [Derived] Rasmussen R, Juhler M, Wetterslev J. Effects of continuous prostacyclin infusion on regional blood flow and cerebral vasospasm following subarachnoid haemorrhage: statistical analysis plan for a randomized controlled trial. Trials. 2014 Jun 14;15:228. doi: 10.1186/1745-6215-15-228. PMID 24929796
- [Derived] Rasmussen R, Wetterslev J, Stavngaard T, Skjoth-Rasmussen J, Grande PO, Olsen NV, Romner B. The effects of continuous prostacyclin infusion on regional blood flow and cerebral vasospasm following subarachnoid haemorrhage: study protocol for a randomised controlled trial. Trials. 2012 Jul 2;13:102. doi: 10.1186/1745-6215-13-102. PMID 22747768